CLINICAL TRIAL: NCT04306328
Title: Functional Evaluation of the Recovery of Prehension in Quadriplegics by Implanted Neural Stimulation
Brief Title: Neural Stimulation for Hand Grasp
Acronym: AGILIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other); NEURINNOV (Unknown); Centre Bouffard Vercelli - USSAP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190280
Record Dates: First submitted 2020-01-31; First posted 2020-03-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Quadriplegia
Keywords: Percutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurostimulation (Experimental)
  Interventions: Device: Neurostimulation

INTERVENTIONS:
Device: Neurostimulation — Implantation of 2 multicontact cuff electrodes in the upper limb of patients with tetraplegia and control of the stimulation by contralateral shoulder movements

SUMMARY:
A selective neural stimulation as the investigators propose allows to stimulate several muscles via a single electrode. Neural stimulation requires less energy for muscle activation. In our approach, 2 electrodes will be implanted above the elbow on the median and radial nerves. This considerably reduces the number of implanted elements and therefore i) the risk of infection, ii) the risk of failure, iii) the surgical risk through minimally invasive surgery.

Our main hypothesis is that multipolar neural electrical stimulation of the median nerve (flexion) and the radial nerve (extension) allows:

* on the one hand, a selective, individualized motor activation (muscle by muscle)
* on the other hand, a synergistic motor activation (association of several muscles) for the purpose of production of functional movements.

DETAILED DESCRIPTION:
Electrical stimulation of the muscles has been used for decades in rehabilitation units specializing in the treatment of spinal cord injuries. It has been shown to be effective in building muscle and preventing muscle atrophy following spinal cord injury (SCI) or stroke. It can also be used to reduce spasticity and above all to promote functionally useful motor control. It is then a Functional Electric Stimulation (FES). In the quadriplegic person marked by a severe motor deficiency of the upper limbs, FES is today the only technique allowing to restore a functional gripping movements in the case where the active muscular resources below the elbows are missing or too weak to allow tendon transfer surgery.

Like "Freehand", all the devices using FES directly stimulate the muscles (surface, intramuscular or epimysial electrodes) and therefore require a high number of internal components with a theoretical risk of infection and greater rejection. since each muscle must be activated via an electrode (up to 12 in the case of "FreeHand"). The investigators propose instead selective neural stimulation as it allows stimulating several muscles via a single electrode. Neural stimulation requires less energy for muscle activation. In our approach, 2 electrodes will be implanted above the elbow on the median and radial nerves. This considerably reduces the number of implanted elements and therefore i) the risk of infection, ii) the risk of failure, iii) the surgical risk thanks to minimally invasive surgery. The procedure consisted of placing a multi-contact cuff electrode around the radial or median nerves and observing the effects of electrical neural stimulation in terms of muscle selectivity, force produced and movement induced. In a previous study, the investigators already proved through acute intra operative testing (under Ethics Committee approval, #NCT03721861) that:

* No failure of the electrodes or of the stimulator was noted.
* For all of the 8 subjects, it was possible to selectively stimulate muscle groups to obtain the opening of the thumb and fingers, or the flexion of the thumb, fingers and obtaining possibly functional grip like the forceps with opposition of the thumb or palmar grip.

A second feasibility study (Ethics committee registration #2016-A00711-50) with 17 quadriplegic patients assessed the subject's ability to use voluntary contractions of sus lesional muscles (EMG recordings in 8 subjects) or voluntary movements of shoulders (inertial recordings in 9 subjects) to control the movements of a robotic hand or the triggering of an electrical surface stimulation of the muscles of the forearm. All of the patients managed to master the proposed interface after a short familiarization period.

On the basis of the results of these two studies, the investigator wish to take an additional step in the development of a gripping assistance device for patients with spinal cord injury:

- by proposing the implantation of two cuff electrodes with percutaneous connection on the arm of quadriplegic people. The electrodes will be kept in place for a period of 1 month before being definitively explanted. An implanted cable will connect the electrodes to an external connector.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patient affiliated to a social security (state medical aid excepted).
* Neurological level ≥ C7
* 18 years old ≤ age ≤ 65 years old,
* complete traumatic injury: defined by an A or B score on the AIS scale. (AIS A or - complete motor deficit under injury. This is an internationally agreed standard for describing spinal cord injury)
* neurological stability (no change in muscle testing) > 6 months,
* post-injury duration > 6 months
* patients without active muscle resources for conventional tendon transfer surgery on the forearm and hand

Exclusion Criteria:

* patient deprived of liberty (by judicial or administrative decision).
* adult patient who is subject to a legal protection measure or unable to express consent
* participation in another ongoing clinical trial
* pregnant or breastfeeding women or women of childbearing age without effective contraception
* spasticity and contractures in flexion or extension of the upper limbs of a destabilizing nature.
* unstable epilepsy with a notion of a epileptic seizure that occurred within the previous 12 months.
* unstable cardiovascular pathology (coronary heart disease, major hypertension, heart failure, etc.).
* infectious pathology under treatment at the inclusion visit
* wearing a pacemaker.
* dermatological problems contraindicating the application of surface electrodes.
* body weight >100 kg
* psychiatric condition and/or history contraindicating participation in research
* any contraindications to anesthesia and/or surgery
* hypersensitivity to low molecular weight heparin (LMWH) or to any of the excipients of the specialty used
* history of immune-mediated heparin-induced thrombocytopenia (HIT) within the last 100 days or presence of circulating antibodies
* clinically significant active bleeding or a condition associated with a high risk of bleeding
* electrical mapping identified as negative during the inclusion visit, i.e. with muscles revealing a rating < 4 MRC for at least one of the extensors (ECRL, ECRB, EDC, EPL) or one of the flexors (FPL, FDS, FDP).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Selectivity index of the configurations which allow an individualized recruitment of the different muscles at D+29 | End of the protocole (day 29)
  Selectivity index of the configurations (active contacts of the electrode and stimulation parameters) which allow an individualized recruitment of the different muscles at D+29 based on the combination of the increase of the Root Mean Square (RMS) value of the Electromyography (EMG) and variation of 10% of the maximum distance covered by the considered segment compared with the rest position.

SECONDARY OUTCOMES:
Motor Capacities Scale (MCS) | Day 29
  The Motor Capacity Scale (MCS) which studies the Key Grip and Grasp sockets in their 3 facets (catching, holding and letting go). MCS should be above 27.
Test n°1 of the 400 Points assessment | Day 29
  functional relevance of neural implantation via the production of 4 movements considered useful: an opening of the 5 fingers, a digito-palmar grip with thumb, a digito-palmar grip without thumb and an end-to-side thumb grip Test No. 1 of the 400 POINTS balance sheet, which brings together the study of 12 hand functions. POINTS score should be above 60.
The rate in % of total tests of grasping objects. | Day 29
  Testing of two methods of autonomous control of the device by the patient. The successful rate in % of total tests of grasping objects. The success rate should be above 80%.
Optimal stimulation strategies obtained for a synergistic functional control | Day 29
  For each movement, the minimum stimulation intensity to produce the movement will be noted. In mA this intensity should be as low as possible. A value above 1.5 mA of failure to obtain the desired movement will be considered as a failed outcome.
The impedance of the electrode contacts. | Day 29
  Assessment of the evolution of the quality of the stimulation over time (stability of the settings and of the tissue / electrode interface). A Impedance of the electrode contacts to assess the state of the contact between the electrode poles and the nerve tissue.
  The state of contact between the electrode poles and the nervous tissue will be evaluated by measuring the impedance of the electrode contacts. This impedance expressed in k ohms, should not be higher than 5. Above this threshold the contact will be considered to be non-functional.
  For each movement, the minimum stimulation intensity (in mA) to initiate the movement should stay below 1.5 mA.
Local skin tolerance | Day 29
  Local skin tolerance assessed by the number of patients with dermatological lesions at the implantation site, of allergic and/or infectious type during the month following implantation. The answer provided daily will be binary yes / no.
Local algological tolerance (1) | Day 29
  Local algological tolerance assessed by number of patients with at least one pain at the implant site, qualified as neuropathic or nociceptive and quantified as > or = 3/10 using a digital analog scale from 0 to 10, during the month following implantation.
Local algological tolerance (2) | Day 29
  Local algological tolerance assessed by average intensity of daily pain

CONTACTS AND LOCATIONS:
Overall Officials: Charles FATTAL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service MPR: USSAP Centre Bouffard-Vercelli, Pôle Santé du, Perpignan, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coste CA, William L, Fonseca L, Hiairrassary A, Andreu D, Geffrier A, Teissier J, Fattal C, Guiraud D. Activating effective functional hand movements in individuals with complete tetraplegia through neural stimulation. Sci Rep. 2022 Oct 6;12(1):16189. doi: 10.1038/s41598-022-19906-x. PMID 36202865